CLINICAL TRIAL: NCT01645904
Title: A Social Media Approach to Improve Genetic Risk Communication Phase I
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Duncan Family Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2012-0418
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Hereditary Diseases
Keywords: Hereditary Diseases; Genetic; Lynch syndrome; Positive or indeterminate test results for Lynch syndrome; Social media; Internet-based program; Questionnaire; Survey; My Family Garden website; Interview; Focus group; Website Analysis and MeasureMent Inventory; WAMMI
MeSH Terms: conditions — Genetic Diseases, Inborn; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Patients participate in audiotaped focus group regarding web-based program, and fill out demographics questionnaire.
  Interventions: Behavioral: Audiotaped Focus Group; Behavioral: Demographic Questionnaire
- Group 2: Patients come to Behavioral Research and Treatment Center (BRTC) at MD Anderson to use initial version of My Family Garden website. Completion of Website Analysis and MeasureMent Inventory (WAMMI), and demographics questionnaires.
  Interventions: Behavioral: Demographic Questionnaire; Behavioral: Audiotaped Interview; Behavioral: WAMMI Inventory
- Group 3: Patients use final version of My Family Garden website, and are interviewed which will be audiotaped. Completion of Website Analysis and MeasureMent Inventory (WAMMI), questionnaire and demographics questionnaire.
  Interventions: Behavioral: Demographic Questionnaire; Behavioral: Audiotaped Interview; Behavioral: WAMMI Inventory

INTERVENTIONS:
Behavioral: Audiotaped Focus Group — Participation in a focus group regarding web-based program designed to improve communication of health and health history information among family members affected by Lynch syndrome.
  Groups: Group 1
Behavioral: Demographic Questionnaire — Complete questions about demographics (age, race, marital status) and medical history. This visit should take about 1 hour to complete.
  Other Names: Surveys
Behavioral: Audiotaped Interview — Group 2: Patients provide feedback regarding initial version of My Family Garden website.
  Group 3: Patients provide feedback regarding final version of My Family Garden website.
  Groups: Group 2; Group 3
Behavioral: WAMMI Inventory — Patients complete Website Analysis and MeasureMent Inventory. This visit should take about 90 minutes to complete.
  Groups: Group 2; Group 3

SUMMARY:
The goal of this research study is to create an internet-based program designed to improve the communication of health and health history information among family members affected by Lynch syndrome.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be assigned to 1 of 3 groups based on when you joined the study.

Group 1:

If you are assigned to Group 1, you will take part in a focus group where you will be asked what you would want in a web-based program designed to improve the communication of health and health history information among family members affected by Lynch syndrome. You will also fill out a questionnaire with questions about your demographics (age, race, marital status) and your medical history. This visit should take about 1 hour to complete.

Group 2:

If you are assigned to Group 2, you will come to the Behavioral Research and Treatment Center (BRTC) at MD Anderson to use the initial version of the My Family Garden website. My Family Garden is designed to teach new ways of communicating about Lynch Syndrome and about other issues related to the disease (such as risks associated with the disease, etc.). You will be instructed on how to use the program by the study staff. After you use the website, you will have an interview where you will provide feedback on your session. You will be asked questions about your feelings about the website and about any possible improvements that could be made to the website. You will also fill out a questionnaire called the Website Analysis and MeasureMent Inventory (WAMMI) which is designed help rate websites. You will also fill out the demographics questionnaire described above.

You will be given the option of completing the WAMMI and demographics questionnaire at the BRTC after your session or at your home. If you choose to complete them at home, you will be provided with a self-addressed, postage-paid envelope so you can mail the questionnaires back to the study staff.

This visit should take about 90 minutes to complete.

Group 3:

If you are assigned to Group 3, you will use the final version of the My Family Garden website. This final version will include changes from the web designers after feedback has been given from the previous groups in this study.

After you use the website, you will have an interview where you will provide feedback on your session. You will be asked questions about your feelings about the website and about any possible improvements that could be made to the website. You will also fill out the WAMMI questionnaire and demographics questionnaire described above.

You will be given the option of coming to the BRTC at MD Anderson to use the My Family Garden computer program or using the program from your home. If you choose to use My Family Garden from your home, you will be given a secure, password-protected hyperlink via e-mail to access the program. You will be instructed on how to use the program by the study staff either in person or over the phone. If you use the program from your home, the study staff will give the interview over the phone. If you complete the questionnaire at your home, you will be provided with a self-addressed, postage-paid envelope so you can mail it back to the study staff.

Whether it is completed at MD Anderson or at home, this visit should last about 90 minutes.

Audiotapes:

All focus groups and interviews will be audiotaped. The audiotapes collected during the course of this study will be stored in locked file cabinets in a locked office and will be destroyed after 5 years.

Length of Study Participation:

Your participation in this study will be over after you have completed the study procedures described above.

This is an investigational study.

Up to 49 participants will be enrolled in this study. All participants will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Able to read and speak english
3. Completion of genetic counseling and testing for a Lynch syndrome mutation
4. Persons with positive (i.e., carrier of Lynch syndrome MMR mutation) as well as indeterminate test results

Exclusion Criteria:

1) None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants recruited from Lynch syndrome families enrolled in the Human Pedigree Analysis Resource (HPAR), MDACC's hereditary cancer registry.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Internet-Based Program Among Lynch Syndrome Family Members | 1 day
  Quantitative analysis include descriptive statistics summarizing participants' demographic and clinical characteristics. Descriptive statistics calculated for each subscale of Website Analysis and MeasureMent Inventory (WAMMI) and for overall measure. Focus groups and interviews transcribed, coded and analyzed. Responses sorted into categorical and conceptual groups, field notes taken during user testing also used to aid in interpretation of interview data.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, MPH, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org